CLINICAL TRIAL: NCT01873768
Title: A Randomized Controlled Trial of Tranexamic Acid and ε-Aminocaproic Acid to Reduce Blood Loss Following Total Knee Arthroplasty
Brief Title: Clinical Efficacy of Tranexamic Acid and ε-Aminocaproic Acid in Reducing Blood Loss Following Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Miller Orthopedic Specialists (Other)
Collaborators: CHI Health Mercy Hospital (Other); Creighton University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOS-16735; MOS1316735 (Other: Miller Orthopedic Specialists)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Tranexamic acid; 6-Aminocaproic Acid; Arthroplasty; Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Antifibrinolytic Agents; Fibrin Modulating Agents; Pharmacologic Actions; Coagulants; Therapeutic Uses
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases | interventions — Tranexamic Acid; Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (TXA) (Active Comparator): 1g in 50ml of saline given over 30 minutes just prior to raising the tourniquet and making the initial incision. A second 1g in 50ml of saline will be infused over 30 minutes beginning at the time of wound closure.
  Interventions: Drug: Tranexamic Acid (TXA)
- ε-Aminocaproic Acid (EACA) (Active Comparator): 7g in 50ml of saline given over 30 minutes just prior to raising the tourniquet and making the initial incision. A second 7g of EACA in 50ml saline will be infused over 30 minutes beginning at the time of wound closure.
  Interventions: Drug: ε-Aminocaproic Acid (EACA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — 1g in 250cc of saline given over 30 minutes just prior to raising the tourniquet and making the initial incision. A second 1g in 250cc of saline will be infused over 30 minutes beginning at the time of wound closure.
  Other Names: Cyklokapron
  Arms: Tranexamic acid (TXA)
Drug: ε-Aminocaproic Acid (EACA) — 7g in 250cc of saline given over 30 minutes just prior to raising the tourniquet and making the initial incision. A second 7g of EACA in 250cc saline will be infused over 30 minutes beginning at the time of wound closure.
  Other Names: Amicar
  Arms: ε-Aminocaproic Acid (EACA)

SUMMARY:
Tranexamic acid (TXA) and ε-aminocaproic acid (EACA) are two drugs shown to limit blood loss following major surgery, from cardiac to orthopedic procedures. Yet compared to tranexamic acid (TXA), research on the clinical impact of ε-aminocaproic acid (EACA) in total knee arthroplasty (TKA) is limited. The primary aim of this study is to determine whether TXA and EACA provide similar blood decreasing effects following TKA or whether one drug provides a superior effect over the other in reducing patients' blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 - 90 years who are scheduled to undergo a unilateral total knee replacement surgery

Exclusion Criteria:

* Non-English speaking individuals
* Individuals with a history of deep vein thrombosis or pulmonary embolism within one year
* Individuals with a history of coagulopathy
* Heart stent within one year
* Pre-operative autologous blood donation
* Unwilling or unable to take Coumadin for deep vein thrombosis (DVT) prophylaxis
* Received nonsteroidal anti-inflammatory drug (NSAID) or platelet antiaggregant treatment within five days prior to surgery
* Pre-operative creatinine greater than 1.5mg/dL

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Transfusion rate | 1.5 to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clifford K Boese, MD, Principal Investigator — Miller Orthopedic Specialists
Locations (1):
- Miller Orthopedic Specialists, Council Bluffs, Iowa, United States